CLINICAL TRIAL: NCT01345058
Title: Open Label Trial of Add on Lacosamide Versus High Dose Monotherapy in Patients With a Seizure Disorder
Brief Title: Add on Lacosamide Versus High Dose Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jong Woo Lee, Associate Neurologist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-001630
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; antiepileptic drug; polytherapy
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lacosamide + Low-Dose Levetiracetam (Experimental): Participants received lacosamide 50 mg twice a day for one week followed by 100 mg twice daily added to low dose levetiracetam ≤1500 mg/day (polytherapy) for 6 months in patients with breakthrough seizures on low-dose levetiracetam.
  Interventions: Drug: lacosamide; Drug: levetiracetam
- Control Group (High-Dose Levetiracetam) (Other): Historical chart review of patients whose dose of levetiracetam was raised to high dose levetiracetam >1500 mg/day (monotherapy) after a breakthrough seizure. No intervention was administered in the study.
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: lacosamide — Lacosamide maximum of 200 mg/day, to be titrated as follows:
  * Week 1: 50 mg twice a day
  * Beginning Week 2: 100 mg twice a day.
  Other Names: Vimpat
  Arms: Lacosamide + Low-Dose Levetiracetam
Drug: levetiracetam — Low dose ≤1500 mg/day, High dose >1500 mg/day

SUMMARY:
This is a study to determine whether a combination of low dose lacosamide and levetiracetam is more effective than high dose levetiracetam in patients who have failed low dose levetiracetam.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 or older
2. Determined to have had at least two partial seizures by an epilepsy specialist, or to have had a single partial seizure with clinical and/or laboratory evidence of a high seizure recurrence risk
3. Monotherapy on levetiracetam less than or equal to 1500 mg/day for at least two weeks
4. Breakthrough seizure while on stable dose (>5 days) of levetiracetam monotherapy regimen, not due to provocative factors (e.g. hypoglycemia, head trauma, missed medications)

Exclusion Criteria:

1. Clinical suspicion of nonepileptic psychogenic seizures or idiopathic generalized epilepsy
2. Pregnant, child-bearing age not using contraception, or breast feeding
3. Medical contraindication to adding lacosamide
4. History of antiepileptic drug (AED) polytherapy
5. Presence of a vagus nerve stimulator
6. Creatinine clearance of less than 50 mL/min
7. Blood pressure instability: pulse <50 or >100, systolic blood pressure (SBP) <50 or >180, clinically significant electrocardiogram (EKG) abnormality
8. History of significant drug rash or anaphylactic reaction with antiepileptic drug
9. Patients with progressive lesions (e.g. brain tumors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2014-02-15 (Actual); Study Completion 2014-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Lee, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Lee JW, Alam J, Llewellyn N, Hurwitz S, Bubrick EB, Sarkis RA, Weisholtz D, Yu H, Putta S, Dworetzky BA, Pennell PB. Open Label Trial of Add on Lacosamide Versus High Dose Levetiracetam Monotherapy in Patients With Breakthrough Seizures. Clin Neuropharmacol. 2016 May-Jun;39(3):128-31. doi: 10.1097/WNF.0000000000000144. PMID 26992155

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam)
Started | 20 | 36
Received Lacosamide | 19 | 0
Completed | 15 | 36
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Participant Reported Increase in Events | 1 | 0
Not completed — Side Effects of Hair Loss and Itchiness | 1 | 0
Not completed — Participant Stopped Taking Study Drug | 1 | 0
Not completed — Participant No-Show at Multiple Visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam) | Total
Number analyzed (Participants) | 20 | 36 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (17.5) | 43.7 (19.8) | 43.4 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 7 | 19 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 36 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Six Month Seizure Freedom
Description: Seizure freedom is defined as having no seizures and was evaluated in the 6 month period after receiving the drug.
Time Frame: 6 Months
Population: All eligible participants. One participant in the Lacosamide + Low-Dose Levetiracetam arm did not receive study drug and is not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam)
Number analyzed (Participants) | 19 | 36
percentage of participants | 47.4 | 41.7
Statistical Analysis 1: Comparison: Lacosamide + Low-Dose Levetiracetam vs Control Group (High-Dose Levetiracetam); Test type: Superiority; p = 0.49, Chi-squared; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.35 to 1.65] — Hazard ratio for seizure occurrence for polytherapy relative to monotherapy

2. Secondary Outcome: Number of Seizure-Free Days
Time Frame: 6 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam)
Number analyzed (Participants) | 19 | 36
days | 118.11 (68.59) | 114.0 (65.06)

3. Secondary Outcome: Time to First Seizure After Therapeutic Dose is Reached
Description: Time in days until the first seizure after the therapeutic dose is reached occurs.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam)
Number analyzed (Participants) | 19 | 36
days | 162.0 [9.0 to 180.0] | 116.5 [6.0 to 180.0]

4. Secondary Outcome: Retention Rate
Description: Retention rate is defined as the percentage of participants who remained on the study drug after study completion.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam)
Number analyzed (Participants) | 19 | 36
percentage of participants | 89 | 80

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence (side effect) in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event that occurs after receiving the drug.
Time Frame: 6 Months
Population: All eligible participants. One participant in the Lacosamide + Low-Dose Levetiracetam arm did not receive study drug and is not included. One participant never confirmed taking the study medication, never followed up, and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam)
Number analyzed (Participants) | 18 | 36
Participants | 11 | 26

ADVERSE EVENTS:
Time Frame: 6 Months
Description: All eligible participants. One participant in the Lacosamide + Low-Dose Levetiracetam arm did not receive study drug and is not included in the analysis. One participant never confirmed taking the study medication, never followed up, and was not included in the analysis.
Arm/Group | Lacosamide + Low-Dose Levetiracetam | Control Group (High-Dose Levetiracetam)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/36
Other Adverse Events (participants affected / at risk) | 11/18 | 26/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide + Low-Dose Levetiracetam (N=18) | Control Group (High-Dose Levetiracetam) (N=36)
Hair Loss (Skin and subcutaneous tissue disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Irritability/depression (Psychiatric disorders) | 1 | 12
Fatigue (General disorders) | 2 | 7
Dizziness (Nervous system disorders) | 1 | 5
Memory/cognitive difficulties/confusion (Psychiatric disorders) | 2 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Decreased libido (Reproductive system and breast disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes